CLINICAL TRIAL: NCT05383391
Title: Knowledge, Practice and Barriers of Foot Self-Care Among Diabetic Patients at Sohag University Hospital
Brief Title: Diabetic Foot Self Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mayyada Elsayed Mohamed Hussien, Mayyada Elsayed Mohamed Hussien, Sohag University
Other Study IDs: Soh-Med-22-05-01
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Foot
Keywords: DPN:Diabetic peripheral neuropathy.; CDC:The center for disease control and prevention .
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study:

Studying patients' knowledge, practice and barriers of foot self-care among diabetic patients attending Sohag University Hospital,.

Objectives:

1. To determine patients' knowledge and practice of foot self-care among diabetic patients attending Sohag University Hospital.
2. To detect barriers of diabetic foot self-care among diabetic patients attending Sohag University Hospital.

Patients and methods:

Place of the study (locality):

Sohag University Hospital at endocrine outpatient clinic .

Type of the study (Study design):

A cross-sectional, descriptive questionnaire based study was designed to evaluate knowledge and practice of diabetic patients regarding foot care.

Period of data collection . 6 months Questionnaires will be distributed among the diabetes mellitus patients in Sohag University Hospital to get the information about the knowledge of the disease among patients. The answer of the questions will be scored with "yes" "no" or I don't "know".

The questionnaire consists of four sections(8):

1. Demographic section .
2. Knowledge related questions regarding foot care .
3. Practice related questions regarding practice of foot care .
4. Barriers to foot self-care . Questionnaire contained 7 questions regarding knowledge of foot care and 12 questions regarding practice of foot care, which was approved and validated by the research committee of faculty of Pharmacy.

DETAILED DESCRIPTION:
Diabetic foot problems are one of the most common chronic complications of diabetes that has a tremendous economic and social impact on individuals, families and on health system as a whole in developing and developed countries.( ) Diabetic foot problems can be prevented through well-coordinated foot care services. Patient education is an important and essential element of any health program for diabetic foot prevention and control. ( ) Diabetic foot problems as one important complication of DM constitute an increasing public health problem and are a leading cause of hospital admission, amputation and mortality in diabetic patients. ( ) Education is the key element in successful management of diabetes, as knowledge about diabetes enables patients to play an active role in effective diabetes self-management.Performing daily foot care routines enables diabetic patients to detect foot abnormalities and injuries earlier, hence reduce or even prevent the risk of foot ulceration effectively. ( ) Diabetic peripheral neuropathy (DPN) is the most common complication of type 2 diabetes mellitus requiring frequent referral for medical or surgical management. ( ) Neuropathy results in loss of sensation in gloves and stocking pattern, which leads to loss of protective sensation to noxious stimuli, such as trauma induced by micro trauma to the skin and bone or trauma caused by stepping on a sharp object or skin injury due to ill fitting shoes.

Moreover, due to modulation of neuro muscular junction the muscles get deprived of their innervations leading to muscle atrophy and foot deformities. Thus, pressures are gradually abnormally distributed on the plantar aspect of the feet, causing an increased forefoot pressure than the rear foot, thereby increasing the risk for ulceration. Initially the situation looks trivial, but the problem posed by DPN in its due course progresses to deep tissue destruction. ( ) The center for disease control and prevention (CDC) reported that complementary foot-care programs including risk assessment, self-foot-care education, metabolic control, and referral to specialists may decrease the risk of amputation by 45%-85%. ( )

ELIGIBILITY:
Inclusion Criteria:

* Known cases of type 2 Diabetes Mellitusaging between 30 and 70 years old.

Exclusion Criteria:

* Emergency ward patients andpatients who were not willing, were excluded from the study.

Patients with toes orfoot amputation, Patients having activefoot ulcers , Patients with cognitive impairment.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Known cases of type 2 Diabetes Mellitusaging between 30 and 70 years old.
  Exclusioncriteria:
  Emergency ward patients andpatients who were not willing, were excluded from the study.
  Patients with toes orfoot amputation, Patients having activefoot ulcers , Patients with cognitive impairment.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Studying patients' knowledge, practice and barriers of foot self-care among diabetic patients attending Sohag University Hospital | 6 months
  A cross-sectional, descriptive questionnaire based study was designed to evaluate knowledge and practice of diabetic patients regarding foot care.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papanas N, Maltezos E. The diabetic foot: a global threat and a huge challenge for Greece. Hippokratia. 2009 Oct;13(4):199-204. PMID 20011082